CLINICAL TRIAL: NCT03486912
Title: A Phase 2B Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of BMS-986036 (PEG-FGF21) in Adults With Nonalcoholic Steatohepatitis (NASH) and Compensated Liver Cirrhosis
Brief Title: A Study of Experimental Medication BMS-986036 in Adults With Nonalcoholic Steatohepatitis (NASH) and Liver Cirrhosis
Acronym: FALCON 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB130-069
Record Dates: First submitted 2018-03-30; First posted 2018-04-03 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hepatic Cirrhosis; Liver Fibrosis; Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986036 Dose Level 1 (Experimental)
  Interventions: Drug: BMS-986036
- BMS-986036 Dose Level 2 (Experimental)
  Interventions: Drug: BMS-986036
- BMS-986036 Dose Level 3 (Experimental)
  Interventions: Drug: BMS-986036
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986036 — Specified dose on specified days.
  Other Names: Pegbelfermin
  Arms: BMS-986036 Dose Level 1; BMS-986036 Dose Level 2; BMS-986036 Dose Level 3
Other: Placebo — Specified dose on specified days.
  Arms: Placebo

SUMMARY:
This is a study of experimental medication BMS-986036 given to adults with Nonalcoholic Steatohepatitis (NASH; the buildup of fat and inflammation in the liver that is not caused by alcohol) and liver cirrhosis (liver damage characterized by normal liver tissue being replaced by scar tissue).

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy performed within 6 months (26 weeks) prior to the screening period. If historical biopsy is not available, a liver biopsy will be performed during the screening period. Biopsy must be consistent with NASH and cirrhosis according to the NASH CRN classification, as assessed by the central reader
* Must be taking anti-diabetic, anti-obesity, or anti-dyslipidemic medications must have been on stable regimens for at least 3 months (12 weeks) (6 weeks for statins) prior to and during the screening period
* Participants taking vitamin E at doses greater than or equal to (>=) 800 IU/day must have been on stable doses for at least 6 months (26 weeks) prior to and during the screening period. Vitamin E treatment (>=800 IU/day) must not have been initiated after the qualifying liver biopsy was performed

Exclusion Criteria:

* Other causes of liver disease (e.g., alcoholic liver disease, hepatitis B virus infection, chronic hepatitis C virus infection [HCV], autoimmune hepatitis, drug-induced hepatotoxicity, Wilson disease, α-1-antitrypsin deficiency, iron overload, and hemochromatosis); participants with HCV sustained viral response (undetectable HCV RNA) for at least 2 years prior to biopsy confirming study eligibility may be eligible
* Current or past history of hepatocellular carcinoma (HCC)
* Past or current evidence of hepatic decompensation (e.g., ascites, variceal bleeding, hepatic encephalopathy and/or spontaneous bacterial peritonitis) or liver transplantation
* Medical history of gastroesophageal varices, except if esophagogastroduodenoscopy [EGD] performed within 12 months prior to the Screening Period has shown <= Grade 1 varices

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (91):
- United States (85):
  - North Alabama Health Research, LLC, Madison, Alabama
  - Local Institution - 0005, Chandler, Arizona
  - Local Institution - 0088, Phoenix, Arizona
  - Local Institution - 0006, Phoenix, Arizona
  - Local Institution - 0090, Tucson, Arizona
  - Kindred Medical Institute for Clinical Trials, Corona, California
  - Local Institution - 0092, Coronado, California
  - Local Institution - 0038, La Jolla, California
  - Local Institution - 0017, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - GastroIntestinal Biosciences, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Kaiser Permanente, Oakland, California
  - Diverse Research Solutions, Oxnard, California
  - Huntington Medical Research Institutes - HMRI Liver Center, Pasadena, California
  - Local Institution - 0020, Pasadena, California
  - Local Institution - 0073, Redwood City, California
  - Local Institution - 0012, Rialto, California
  - Local Institution - 0089, San Clemente, California
  - Local Institution, San Diego, California
  - Local Institution - 0014, San Diego, California
  - Local Institution - 0068, San Francisco, California
  - Local Institution - 0042, Bridgeport, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution - 0079, Coral Gables, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Clinical Research of Homestead, Homestead, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Local Institution - 0001, Lakewood Rch, Florida
  - Local Institution - 0003, Miami, Florida
  - A+ Research, Miami, Florida
  - IMIC Research, Miami, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Local Institution - 0081, Orlando, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution - 0108, Marietta, Georgia
  - Tandem Clinical Research, Marrero, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Local Institution - 0026, New Orleans, Louisiana
  - Local Institution - 0010, Baltimore, Maryland
  - Local Institution - 0058, Catonsville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Local Institution - 0031, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - University at Buffalo, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Local Institution - 0036, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Local Institution - 0067, Butner, North Carolina
  - Local Institution - 0064, Charlotte, North Carolina
  - Northeast GI Research Division, Concord, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Local Institution - 0009, Philadelphia, Pennsylvania
  - Local Institution - 0004, Pittsburgh, Pennsylvania
  - Local Institution, Chattanooga, Tennessee
  - Local Institution - 0046, Germantown, Tennessee
  - Local Institution - 0041, Hermitage, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Local Institution - 0066, Austin, Texas
  - Local Institution - 0051, Dallas, Texas
  - Local Institution - 0053, Dallas, Texas
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0084, Fort Worth, Texas
  - Local Institution - 0002, Houston, Texas
  - Local Institution - 0057, Houston, Texas
  - Local Institution - 0063, Houston, Texas
  - Local Institution - 0028, San Antonio, Texas
  - Local Institution - 0011, San Antonio, Texas
  - Local Institution - 0102, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Gastroenterology Associates, PC, Manassas, Virginia
  - Local Institution - 0069, Norfolk, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Local Institution - 0077, Richmond, Virginia
  - Local Institution - 0050, Richmond, Virginia
- Japan (6):
  - Kurume University Hospital, Kurume, Fukuoka
  - Local Institution - 0055, Yokohama, Kanagawa
  - Local Institution - 0072, Kashihara, Nara
  - Toranomon Hospital, Minato, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Fukushima Medical University Hospital, Fukushima

REFERENCES:
- [Derived] Abdelmalek MF, Sanyal AJ, Nakajima A, Neuschwander-Tetri BA, Goodman ZD, Lawitz EJ, Harrison SA, Jacobson IM, Imajo K, Gunn N, Halegoua-DeMarzio D, Akahane T, Boone B, Yamaguchi M, Chatterjee A, Tirucherai GS, Shevell DE, Du S, Charles ED, Loomba R. Pegbelfermin in Patients With Nonalcoholic Steatohepatitis and Compensated Cirrhosis (FALCON 2): A Randomized Phase 2b Study. Clin Gastroenterol Hepatol. 2024 Jan;22(1):113-123.e9. doi: 10.1016/j.cgh.2023.04.012. Epub 2023 Apr 23. PMID 37088458
- [Derived] Abdelmalek MF, Charles ED, Sanyal AJ, Harrison SA, Neuschwander-Tetri BA, Goodman Z, Ehman RA, Karsdal M, Nakajima A, Du S, Tirucherai GS, Klinger GH, Mora J, Yamaguchi M, Shevell DE, Loomba R. The FALCON program: Two phase 2b randomized, double-blind, placebo-controlled studies to assess the efficacy and safety of pegbelfermin in the treatment of patients with nonalcoholic steatohepatitis and bridging fibrosis or compensated cirrhosis. Contemp Clin Trials. 2021 May;104:106335. doi: 10.1016/j.cct.2021.106335. Epub 2021 Feb 28. PMID 33657443
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986036 10 mg: BMS-986036 10 mg administered subcutaneously once weekly
- BMS-986036 20 mg: BMS-986036 20 mg administered subcutaneously once weekly
- BMS-986036 40 mg: BMS-986036 40 mg administered subcutaneously once weekly
- Placebo: Placebo matching BMS-986036 administered subcutaneously once weekly
Period: Randomized (Pre-Treatment)
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Started | 39 | 38 | 39 | 39
Completed (Moved to treatment period) | 39 | 37 | 39 | 39
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Treatment Period
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Started | 39 | 37 | 39 | 39
Completed | 35 | 31 | 34 | 34
Not Completed | 4 | 6 | 5 | 5
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 2
Not completed — Other Reasons | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 39 | 39 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 30 | 25 | 112
  >=65 years | 12 | 8 | 9 | 14 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 21 | 24 | 99
  Male | 11 | 12 | 18 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 7 | 11 | 37
  Not Hispanic or Latino | 25 | 30 | 31 | 28 | 114
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 4 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 30 | 31 | 34 | 33 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Achieve a ≥ 1-Stage Improvement in Fibrosis Without Worsening of Nonalcoholic Steatohepatitis (NASH) at Week 48
Description: An improvement in fibrosis is defined as a decrease of fibrosis by ≥1-stage in the NASH Clinical Research Network (CRN) Fibrosis Score at week 48 in liver biopsy. Worsening of NASH is defined as an increase of the nonalcoholic fatty liver disease activity score (NAS) by ≥ 1-stage.
  Worsening of NASH is defined as an increase of the nonalcoholic fatty liver disease (NAFLD) Activity Score (NAS) by ≥1 point. Worsening of fibrosis is defined as an increase of fibrosis by ≥1 point as determined by the NASH CRN Fibrosis Score.
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 28.2 | 24.3 | 28.2 | 30.8
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.773, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.30 to 2.62]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.544, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.23 to 2.23]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.811, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.30 to 2.62]

2. Secondary Outcome: The Percentage of Participants Who Achieve a ≥ 1-Stage Improvement in Ishak Fibrosis Score at Week 48
Description: An improvement in Ishak fibrosis is defined as a decrease of fibrosis by ≥ 1-stage in the Ishak fibrosis score at week 48 in liver biopsy. ISHAKs uses a 0-6 scale: 1: centrilobular pericellular fibrosis, 2: centrilobular and periportal fibrosis, 3: bridging fibrosis (few bridges), 4: bridging fibrosis (many bridges), 5: early or incomplete cirrhosis, 6: established or advanced cirrhosis.
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 38.5 | 32.4 | 33.3 | 35.9
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.836, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.40 to 3.09]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.763, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.30 to 2.46]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.821, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.32 to 2.51]

3. Secondary Outcome: The Percentage of Participants With Improvement in Fibrosis Without Worsening of Nonalcoholic Steatohepatitis (NASH) or NASH Improvement at Week 48
Description: The percentage of participants who achieved a ≥1-stage improvement in fibrosis without worsening of NASH or NASH improvement with no worsening of fibrosis at week 48 in liver biopsy. Improvement in fibrosis is defined by the NASH Clinical Research Network (CRN) Fibrosis Score. Improvement in NASH is defined by a ≥2-stage decrease in the nonalcoholic fatty liver disease activity score (NAS). NASH CRN Fibrosis is staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 33.3 | 40.5 | 35.9 | 30.8
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.837, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.39 to 3.25]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.359, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.54 to 4.40]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.627, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.44 to 3.61]

4. Secondary Outcome: The Percentage of Participants Who Achieved >=1 Point Improvement in Fibrosis at Week 48
Description: An improvement in fibrosis is defined as a decrease of ≥ 1-stage in the non-alcoholic steatohepatitis clinical research network (NASH CRN) Fibrosis Score at week 48 in liver biopsy. NASH CRN Fibrosis is staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 35.9 | 29.7 | 28.2 | 33.3
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.864, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.40 to 3.16]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.743, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.29 to 2.49]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.630, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.27 to 2.29]

5. Secondary Outcome: The Percentage of Participants With Any Improvement in Collagen Proportionate Area (CPA) at Week 48
Description: An improvement in CPA is defined as any decrease in CPA at week 48 in liver biopsy.
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 61.8 | 54.2 | 41.9 | 53.1
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.477, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.48 to 4.25]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.814, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.32 to 3.44]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.367, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.21 to 1.93]

6. Secondary Outcome: The Percentage of Participants With Nonalcoholic Steatohepatitis (NASH) Resolution at Week 48
Description: NASH resolution defined by the nonalcoholic fatty liver disease activity score (NAS) component of ballooning = 0 and inflammation = 0-1 at week 48 in liver biopsy. Ballooning = 0 (none) inflammation = 0 (none) - 1 (Grade <2).
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 2.6 | 5.4 | 2.6 | 0.0
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.309, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.146, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.317, Cochran-Mantel-Haenszel

7. Secondary Outcome: The Percentage of Participants With Nonalcoholic Steatohepatitis (NASH) Improvement at Week 48
Description: The percentage of participants with NASH improvement at week 48 in liver biopsy. NASH improvement is defined as a reduction of nonalcoholic fatty liver disease activity score (NAS) by ≥ 2 points with contribution from > 1 NAS component. The NASH CRN system assesses liver biopsies for degree of steatosis (0-3), lobular inflammation (0-3), hepatocellular ballooning (0-2), and fibrosis (0-4). The 3 categories are added together in an unweighted fashion to determine the NAS, which ranges from 0 to 8.
Time Frame: From first dose to 48 weeks after first dose
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
Number analyzed (Participants) | 39 | 37 | 39 | 39
Percentage of Participants | 15.4 | 24.3 | 12.8 | 2.6
Statistical Analysis 1: Comparison: BMS-986036 10 mg vs Placebo; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.91, 95% CI 2-sided [0.76 to 325.97]
Statistical Analysis 2: Comparison: BMS-986036 20 mg vs Placebo; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 12.21, 95% CI 2-sided [1.50 to 549.08]
Statistical Analysis 3: Comparison: BMS-986036 40 mg vs Placebo; Test type: Superiority; p = 0.087, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.59, 95% CI 2-sided [0.57 to 271.11]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from their randomization until the study was completed (up to approximately 39 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 52 weeks).
Description: All-cause mortality was assessed for all randomized participants. SAEs and Other AEs were assessed for all treated participants.
Arm/Group | BMS-986036 10 mg | BMS-986036 20 mg | BMS-986036 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/39 | 0/38 | 0/39 | 1/39
Serious Adverse Events (participants affected / at risk) | 7/39 | 7/37 | 8/39 | 3/39
Other Adverse Events (participants affected / at risk) | 27/39 | 36/37 | 29/39 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986036 10 mg (N=39) | BMS-986036 20 mg (N=37) | BMS-986036 40 mg (N=39) | Placebo (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986036 10 mg (N=39) | BMS-986036 20 mg (N=37) | BMS-986036 40 mg (N=39) | Placebo (N=39)
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 6 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 16 | 11 | 6
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 3 | 6 | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 11 | 7 | 5
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Fatigue (General disorders) | 1 | 6 | 1 | 1
Injection site bruising (General disorders) | 2 | 7 | 3 | 4
Injection site erythema (General disorders) | 1 | 1 | 5 | 2
Injection site pain (General disorders) | 2 | 2 | 3 | 1
Injection site reaction (General disorders) | 0 | 2 | 2 | 0
Injection site swelling (General disorders) | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 2 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 2
Acute sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 4 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 3
Furuncle (Infections and infestations) | 0 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2 | 2
Influenza (Infections and infestations) | 1 | 2 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 5 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 5 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 2 | 4 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 2
Vitamin D decreased (Investigations) | 0 | 1 | 2 | 0
Weight increased (Investigations) | 2 | 0 | 2 | 0
White blood cells urine positive (Investigations) | 0 | 3 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 6 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 2 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 4 | 2 | 5
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03486912/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03486912/SAP_001.pdf